CLINICAL TRIAL: NCT04845659
Title: Treatment With Avatrombopaq in Patients With Cirrhosis Undergoing Small Invasive Procedure: A Prospective Case Series
Brief Title: Avatrombopaq In Patients With Cirrhosis
Acronym: AIPAC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Christian Snitkjær, M.B., Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AIPAC21
Record Dates: First submitted 2021-04-11; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Thrombocytopenia; Drugs; Cirrhosis, Liver; Procedural Bleeding
Keywords: Cirrhosis; Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia; Liver Cirrhosis; Fibrosis | interventions — avatrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Avatrombopaq administration
  Interventions: Drug: Doptelet Pill

INTERVENTIONS:
Drug: Doptelet Pill — 40 mg or 60 mg Doptelet orally 10-13 days before planned procedure.

SUMMARY:
Thrombocytopenia is a frequent issue in patients with cirrhosis undergoing various types of procedures (e.g. liver biopsy, endoscopy and minor surgical interventions). Thrombocytopenia < 50*10^9/L increases the risk of perioperative and postoperative bleedning and might prevent patients with cirrhosis to undergo important procedures. Doptelet is a small molecular trombopoetin agonist, which results in proliferation and differentiation of megakaryocytes in the bone marrow resulting in increased levels of thrombocytes. It is given orally as a pill and is used to increase platelet count in patients with severe thrombocytopenia (< 50*10^9/L) and cirrhosis and thus not to normalize platelet count. This study investigates the safety and efficacy of Doptelet in patients with cirrhosis and thrombocytopenia (< 50*10^9/L) undergoing minor procedures like Transjugular Adjusted Liver Biopsy (TJALB) and gastroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age: >17 years and ≤80 years
* ASA I-III
* Patients who read, understood and signed informed consent.
* Patients with a diagnosis of cirrhosis
* Thrombocytopenia <50*109
* The patient is scheduled for one of the following procedures: Transjugular Adjusted Liver Biopsy (TJALB), gastroscopy or percutan paracentesis of ascites in the following month.

Exclusion Criteria:

* Patients who do not speak and understand Danish.
* Patients who cannot cooperate within the trial.
* Patients who did not sign an informed consent regardless of the cause.
* Active drug abuse - to the discretion of the investigator.
* Thrombocytes >50*10^9
* Patients with hereditary trombolic diseases (e.g. Factor V Leiden, antithrombin deficiency, protein S and C deficiency, prothrombin G202110A mutation).
* INR > 1,7
* Ongoing infection verified by blood culture, clinical examination, and acute phase reactants (e.g. CRP)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 3 months postprocedural
  Mortality, bleedning, blood clots, readmission, reoperation

IPD SHARING:
Plan to Share IPD: No